CLINICAL TRIAL: NCT03118518
Title: STOP AF First: Cryoballoon Catheter Ablation in an Antiarrhythmic Drug Naive Paroxysmal Atrial Fibrillation
Acronym: STOP AF First
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT16012AFS001
Record Dates: First submitted 2017-04-04; First posted 2017-04-18 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation New Onset
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery; Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Anti-arrhythmic drug (Active Comparator)
  Interventions: Drug: Antiarrhythmic drug
- Cryoablation (Experimental)
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Pulmonary vein isolation via ablation with cryoballoon catheter
  Other Names: ArcticFront Advance Cardiac CryoAblation Catheter
  Arms: Cryoablation
Drug: Antiarrhythmic drug — Antiarrhythmic drug initiation
  Arms: Anti-arrhythmic drug

SUMMARY:
To provide data demonstrating the safety and effectiveness of the Arctic Front Advance™ Cardiac CryoAblation Catheter for the treatment of recurrent symptomatic paroxysmal atrial fibrillation, without the requirement that the subjects be drug refractory.

DETAILED DESCRIPTION:
Subjects with paroxysmal atrial fibrillation with no history of treatment with anti-arrhythmic drugs are randomized 1:1 to either an anti-arrhythmic drug or pulmonary vein isolation using the cryoballoon catheter.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of symptomatic paroxysmal AF with the following documentation: (1) physician's note indicating recurrent self- terminating AF or paroxysmal AF; and (2) any ECG documented AF within 6 months prior to enrollment.
* Age 18-80

Exclusion Criteria:

* History of AF treatment with class I or III antiarrhythmic drug, including sotalol, with the intention to prevent an AF recurrence. However, patients pretreated with above AAD for less than 7 days with the intention to convert an AF episode are allowed.
* Prior persistent AF (cardioversion after 48 hours or continuous AF that is sustained >7 days)
* Left atrial diameter greater than 5.0 cm
* Prior left atrial ablation or left atrial surgical procedure
* Presence or likely implant of a permanent pacemaker, biventricular pacemaker, loop recorder, or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
* Body mass index (BMI) >35 kg/m2
* Presence of any pulmonary vein stents
* Known presence of any pre-existing pulmonary vein stenosis
* Pre-existing hemidiaphragmatic paralysis
* Presence of any cardiac valve prosthesis
* Moderate or severe mitral valve regurgitation or stenosis
* Any cardiac surgery, myocardial infarction, percutaneous coronary intervention/ percutaneous transluminal coronary angioplasty or coronary artery stenting which occurred during the 90 day interval preceding the date the subject signed the Informed Consent Form
* Unstable angina
* New York Heart Association (NYHA) class III or IV congestive heart failure and/or known left ventricular ejection fraction (LVEF) less than 45%
* Diagnosis of primary pulmonary hypertension
* Rheumatic heart disease
* Thrombocytosis, thrombocytopenia
* Contraindication to anticoagulation therapy
* Active systemic infection
* Hypertrophic cardiomyopathy
* Cryoglobulinemia
* Known reversible causes of AF, including but not limited to uncontrolled hyperthyroidism, obstructive sleep apnea, and acute alcohol toxicity.
* Any cerebral ischemic event (strokes or transient ischemic attacks) which occurred during the 180 day interval preceding the date the subject signed the Informed Consent Form, or any known unresolved complications from previous stroke/transient ischemic attack
* Existing thrombus
* Pregnancy
* Patient with life expectancy that makes it unlikely 12 months of follow-up will be completed.
* Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of this study not pre-approved by Medtronic
* Patients with contraindications to a Holter monitor
* Unwilling or unable to comply fully with study procedures and follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 225 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Wazni, MD, Principal Investigator — The Cleveland Clinic; Gopi Dandamudi, MD, Principal Investigator — Franciscan Heart & Vascular Associates at St. Joseph; Steve Nissen, MD, Principal Investigator — The Cleveland Clinic
Locations (24):
- United States (24):
  - Grandview Medical Center, Birmingham, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Hoag Hospital Newport Beach, Newport Beach, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tallahassee Research Institute Inc, Tallahassee, Florida
  - BayCare Medical Group Cardiology, Tampa, Florida
  - Wellstar Research Institute, Marietta, Georgia
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Our Lady of the Lake Office of Research, Baton Rouge, Louisiana
  - Southcoast Health System, New Bedford, Massachusetts
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - HealthEast Saint Josephs Hospital, Saint Paul, Minnesota
  - Bryan Heart, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Health, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrade JG, Moss JWE, Kuniss M, Sadri H, Wazni O, Sale A, Ismyrloglou E, Chierchia GB, Kaplon R, Mealing S, Bainbridge J, Bromilow T, Lane E, Khaykin Y. The Cost-Effectiveness of First-Line Cryoablation vs First-Line Antiarrhythmic Drugs in Canadian Patients With Paroxysmal Atrial Fibrillation. Can J Cardiol. 2024 Apr;40(4):576-584. doi: 10.1016/j.cjca.2023.11.019. Epub 2023 Nov 23. PMID 38007219
- [Derived] Wazni OM, Dandamudi G, Sood N, Hoyt R, Tyler J, Durrani S, Niebauer M, Makati K, Halperin B, Gauri A, Morales G, Shao M, Cerkvenik J, Kaplon RE, Nissen SE; STOP AF First Trial Investigators. Cryoballoon Ablation as Initial Therapy for Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):316-324. doi: 10.1056/NEJMoa2029554. Epub 2020 Nov 16. PMID 33197158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first enrollment in the STOP AF First study occurred in the United States on 23-JUN-2017. The final enrollment occurred on 13-MAY-2019.
Pre-assignment Details: Of 225 enrolled participants, 210 met inclusion criteria and were randomized to treatment. Of the 15 who exited prior to randomization: 11 did not meet inclusion/exclusion criteria, 2 withdrew, 1 was lost to follow-up and 1 had study enrollment close prior to randomization.
Groups:
- Subjects Randomized to Cryoballoon Catheter Ablation: Subjects Randomized to Cryoballoon Catheter Ablation.
- Subjects Randomized to Antiarrhythmic Drug Therapy: Subjects Randomized to Antiarrhythmic Drug Therapy.
Period: Overall Study
Arm/Group | Subjects Randomized to Cryoballoon Catheter Ablation | Subjects Randomized to Antiarrhythmic Drug Therapy
Started | 108 | 102
Subject Treated According to Randomization Assignment | 104 | 99
Completed | 102 | 91
Not Completed | 6 | 11
Not completed — Early Exit after treatment | 2 | 8
Not completed — Early Exit after randomization but prior to treatment | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects Treated With Cryoballoon Catheter Ablation as Randomized: Subjects Treated with Cryoballoon Catheter Ablation as Randomized.
- Subjects Treated With Antiarrhythmic Drug Initiation: Subjects Treated with Antiarrhythmic Drug Initiation.
- Total: Total of all reporting groups
Arm/Group | Subjects Treated With Cryoballoon Catheter Ablation as Randomized | Subjects Treated With Antiarrhythmic Drug Initiation | Total
Number analyzed (Participants) | 104 | 99 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 49 | 108
  >=65 years | 45 | 50 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.2) | 61.6 (11.2) | 61.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 63 | 57 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 97 | 91 | 188
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 94 | 91 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 104 | 99 | 203

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success at 12 Months After Antiarrhythmic Drug (AAD) Initiation or Ablation Utilizing the Arctic Front Advance™ Cardiac CryoAblation Catheter.
Description: Treatment success after AAD initiation (control arm) or pulmonary vein isolation ablation procedure utilizing the Arctic Front Advance™ Cardiac CryoAblation Catheter (treatment arm). Treatment success is the opposite of treatment failure. Treatment failure was defined as any of the following:
  * Acute procedural failure (treatment arm only).
  * Documented AF/AT/AFL on ambulatory monitoring/12-lead ECG after the 90-day post-ablation blanking period (treatment)/AAD optimization period (control arm). Minimum of 30 seconds on ambulatory monitoring or 10 seconds on 12-lead ECG.
  * Any subsequent AF surgery or ablation in the left atrium.
  * Any subsequent cardioversion after the 90-day post-ablation blanking period (treatment)/AAD optimization period (control arm).
  * Class I or III antiarrhythmic drug (or sotalol) use after the 90-day blanking period (treatment arm only).
Time Frame: Randomization to 12 months
Population: Subjects who were received the treatment they were randomized to (modified intent to treat).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Treated With Cryoballoon Catheter Ablation as Randomized | Subjects Treated With Antiarrhythmic Drug Initiation
Number analyzed (Participants) | 104 | 99
percentage of participants | 73.7 [64.0 to 81.2] | 45.0 [34.6 to 54.7]

2. Primary Outcome: Primary Safety Endpoint - Rate of Composite List of Serious Adverse Events.
Description: Measured by rate of composite list of serious adverse events in cryoablation-treated as randomized arm.
  Includes:
  * TIA within 7 days
  * Cerebrovascular accident within 7 days
  * Major bleed that requires transfusion or results in a 20% or greater fall in hematocrit (HCT) within 7 days
  * Development of a significant pericardial effusion within 30 days. (One that results in hemodynamic compromise, requires elective or urgent pericardiocentesis, or results in a 1-cm or more pericardial effusion as documented by echocardiography).
  * Symptomatic PV stenosis within 12 months; accompanied by one of the following: 50%-75% reduction in diameter of the pulmonary vein, with symptoms not explained by other conditions; OR >75% reduction in diameter of the pulmonary vein
  * MI within 7 days
  * PNI unresolved at 12 months
  * AE fistula within 12 months
  * Major vascular complication that requires intervention, prolongs hospital stay, or requires hospital admission (within 7 days).
Time Frame: Randomization to 12 months
Population: Subjects who were cryoablation-treated as randomized (as was pre-specified in both the protocol and Statistical Analysis Plan)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Treated With Cryoballoon Catheter Ablation as Randomized
Number analyzed (Participants) | 104
percentage of participants | 1.92 [0.48 to 7.47]

3. Secondary Outcome: Quality of Life Scores at Baseline Compared to 12 Months
Description: There are two hypotheses tested in the objective, with separate hypothesis tests for (1) the difference in composite scores from the AFEQT questionnaire taken at baseline and 12 month visits, and (2) for the difference in composite scores for the EQ-5D questionnaire taken at baseline and 12-month visits.
  Composite AFEQT score is on a scale of zero to one hundred. Higher scores are better.
  Composite EQ-5D score is on a scale of zero to one. Higher scores are better.
Time Frame: Baseline and 12 Months
Population: Subjects treated with cryoballoon catheter ablation as randomized (as was pre-specified in both the protocol and Statistical Analysis Plan) and who had QOL score available at both baseline and 12 month time points.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Subjects Treated With Cryoballoon Catheter Ablation as Randomized
Number analyzed (Participants) | 99
Score on a scale
  AFEQT composite score (change from baseline to 12 months) | 33.3 [29.1 to 37.5]
  Composite EQ-5D score (change from baseline to 12 months) | 0.04 [0.01 to 0.06]

4. Secondary Outcome: Healthcare Utilization
Description: Compare health care utilization between the treatment and control arms. There are two hypotheses tested in the objective, with separate hypothesis tests for: (1) the rate of total health care utilization events (cardiovascular-related hospitalizations, emergency room visits, or unscheduled office visits) over 12 months shown as freedom from cardiovascular health care utilization by treatment arm, and (2) freedom from cardioversions (electrical or pharmacological) over 12 months by treatment arm.
Time Frame: Initial treatment through 12 months.
Population: All subjects treated as randomized (mITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects Treated With Cryoballoon Catheter Ablation as Randomized | Subjects Treated With Antiarrhythmic Drug Initiation
Number analyzed (Participants) | 104 | 99
percentage of participants
  Freedom from Cardiovascular health care utilization. | 69.9 [60.0 to 77.8] | 53.5 [42.8 to 63.1]
  Freedom from Cardioversion | 97.1 [91.3 to 99.1] | 92.4 [84.8 to 96.3]

ADVERSE EVENTS:
Time Frame: During or after treatment initiation through study completion (12 months visit).
Description: Adverse events occurring during the study were continuously monitored and collected.
  The following adverse events were collected starting at the time subjects signed the Informed Consent Form through the duration of the subject's participation in the study:
  * All procedure related AEs
  * All cryoablation system related AEs
  * All AAD related AEs
  * All cardiovascular related AEs
  * All Serious Adverse Events (SAEs), regardless of relatedness
Groups:
- Randomized and Treated With Cryoablation: Subjects Treated with Cryoballoon Catheter Ablation as Randomized.
- Randomized and Treated With Antiarrhythmic Drugs: Subjects Treated with Antiarrhythmic Drug Initiation as Randomized
Arm/Group | Randomized and Treated With Cryoablation | Randomized and Treated With Antiarrhythmic Drugs
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/99
Serious Adverse Events (participants affected / at risk) | 16/104 | 14/99
Other Adverse Events (participants affected / at risk) | 8/104 | 16/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized and Treated With Cryoablation (N=104) | Randomized and Treated With Antiarrhythmic Drugs (N=99)
Acute myocardial infarction (Cardiac disorders) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac sarcoidosis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Stenosis (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Presyncope (Vascular disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized and Treated With Cryoablation (N=104) | Randomized and Treated With Antiarrhythmic Drugs (N=99)
Atrial fibrillation (Cardiac disorders) | 8 (12) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Version 4 (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03118518/Prot_004.pdf
  • Study Protocol: Version 5 (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03118518/Prot_005.pdf
  • Study Protocol: Version 6 (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03118518/Prot_006.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03118518/SAP_007.pdf